CLINICAL TRIAL: NCT00358215
Title: A Double-blind, Randomized, Placebo-controlled, Multicenter Study to Assess the Efficacy and Safety of Darbepoetin Alfa Treatment on Mortality and Morbidity in Heart Failure (HF) Subjects With Symptomatic Left Ventricular Systolic Dysfunction and Anemia
Brief Title: RED-HF™ Trial - Reduction of Events With Darbepoetin Alfa in Heart Failure Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20050222; RED-HF™ Trial
Record Dates: First submitted 2006-07-27; First posted 2006-07-31 (Estimated); Results first posted 2013-12-13 (Estimated); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Heart Failure; Anemia; Cardiovascular Disease; Ventricular Dysfunction; Congestive Heart Failure
Keywords: Survival study; morbidity and mortality; heart failure hospitalization; all-cause death; patient-reported outcomes; Kansas City Cardiomyopathy questionnaire; anemia treatment
MeSH Terms: conditions — Heart Failure; Anemia; Cardiovascular Diseases; Ventricular Dysfunction | interventions — Darbepoetin alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Darbepoetin alfa (Experimental): Starting dose of 0.75 µg/kg subcutaneously every 2 weeks until hemoglobin concentrations reach 13.0 g/dL on 2 consecutive visits, then monthly dosing, titrated to achieve hemoglobin target of 13.0 g/dL, not to exceed 14.5 g/dL.
  Interventions: Drug: Darbepoetin alfa
- Placebo (Placebo Comparator): Participants received dose and administration schedule (every 2 weeks or once a month) changes that simulated the changes for participants receiving darbepoetin alfa.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Darbepoetin alfa — Administered by subcutaneous injection
  Other Names: Aranesp®
  Arms: Darbepoetin alfa
Drug: Placebo — Placebo subcutaneous injection
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine the efficacy of treatment of anemia with darbepoetin alfa compared to placebo on the composite of time to death from any cause or first hospital admission for worsening heart failure in patients with symptomatic left ventricular systolic dysfunction and anemia.

DETAILED DESCRIPTION:
Several epidemiological studies have demonstrated an association between HF and anemia and correlation of increased risk for mortality and hospitalization with low hemoglobin in patients with HF. Earlier single-center interventional studies suggest that meaningful clinical benefits may be achieved by raising hemoglobin concentration in patients with symptomatic HF and anemia. Data from Amgen's completed phase 2 multi-center studies support this hypothesis and show that darbepoetin alfa is well tolerated in patients with symptomatic left ventricular systolic dysfunction and anemia and effectively raises hemoglobin. The pivotal phase 3 Study 20050222 RED-HF Trial is evaluating the effect of treatment with darbepoetin alfa on the composite risk of all-cause mortality or hospitalization for worsening HF in patients with symptomatic left ventricular systolic dysfunction and anemia. This study also evaluates the effect of darbepoetin alfa treatment on all-cause death, on cardiovascular death or hospitalization for worsening HF, and on patient-reported quality-of-life outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure of at least 3 months duration and of New York Heart Association (NYHA) class II, III, or IV
* hemoglobin between 9.0 g/dL and 12.0 g/dL
* left ventricular ejection fraction equal to or less than 40%

Exclusion Criteria:

* Transferrin saturation (Tsat) < 15%
* Blood pressure > 160/100 mm Hg
* Heart failure primarily due to valvular heart disease or clinically significant valvular heart disease that might lead to surgical correction within 12 months of randomization
* Recipient of a major organ transplant or receiving renal replacement therapy
* Serum creatinine > 3.0 mg/dL (> 265 µmol/L)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2278 (Actual)
Dates: Start 2006-06-01 (Actual); Primary Completion 2012-10-11 (Actual); Study Completion 2012-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (575):
- United States (198):
  - Research Site, Birmingham, Alabama
  - Research Site, Huntsville, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Gilbert, Arizona
  - Research Site, Mesa, Arizona
  - Research Site, Scottsdale, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Anaheim, California
  - Research Site, Buena Park, California
  - Research Site, Corona, California
  - Research Site, Culver City, California
  - Research Site, Downey, California
  - Research Site, La Jolla, California
  - Research Site, Lancaster, California
  - Research Site, Larkspur, California
  - Research Site, Loma Linda, California
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Modesto, California
  - Research Site, Oakland, California
  - Research Site, Pasadena, California
  - Research Site, Redondo Beach, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, San Francisco, California
  - Research Site, Santa Monica, California
  - Research Site, Santa Rosa, California
  - Research Site, Sylmar, California
  - Research Site, Walnut Creek, California
  - Research Site, Westlake Village, California
  - Research Site, Aurora, Colorado
  - Research Site, Colorado Springs, Colorado
  - Research Site, Denver, Colorado
  - Research Site, Littleton, Colorado
  - Research Site, Loveland, Colorado
  - Research Site, Bridgeport, Connecticut
  - Research Site, Fairfield, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Jacksonville, Florida
  - Research Site, Jacksonville Beach, Florida
  - Research Site, Jupiter, Florida
  - Research Site, Melbourne, Florida
  - Research Site, Miami, Florida
  - Research Site, Miami Beach, Florida
  - Research Site, Orlando, Florida
  - Research Site, Port Charlotte, Florida
  - Research Site, Safety Harbor, Florida
  - Research Site, Sarasota, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Tamarac, Florida
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Augusta, Georgia
  - Research Site, Covington, Georgia
  - Research Site, Rome, Georgia
  - Research Site, Meridian, Idaho
  - Research Site, Chicago, Illinois
  - Research Site, Elk Grove Village, Illinois
  - Research Site, Evanston, Illinois
  - Research Site, Hinsdale, Illinois
  - Research Site, Maywood, Illinois
  - Research Site, Melrose Park, Illinois
  - Research Site, Oak Lawn, Illinois
  - Research Site, Oakbrook Terrace, Illinois
  - Research Site, Peoria, Illinois
  - Research Site, Rockford, Illinois
  - Research Site, Springfield, Illinois
  - Research Site, Anderson, Indiana
  - Research Site, Fort Wayne, Indiana
  - Research Site, Indianapolis, Indiana
  - Research Site, Jeffersonville, Indiana
  - Research Site, Valparaiso, Indiana
  - Research Site, Des Moines, Iowa
  - Research Site, Iowa City, Iowa
  - Research Site, Kansas City, Kansas
  - Research Site, Olathe, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Louisville, Kentucky
  - Research Site, Madisonville, Kentucky
  - Research Site, Alexandria, Louisiana
  - Research Site, Covington, Louisiana
  - Research Site, Lake Charles, Louisiana
  - Research Site, Marrero, Louisiana
  - Research Site, Slidell, Louisiana
  - Research Site, South Portland, Maine
  - Research Site, Annapolis, Maryland
  - Research Site, Baltimore, Maryland
  - Research Site, Salisbury, Maryland
  - Research Site, Ayer, Massachusetts
  - Research Site, Boston, Massachusetts
  - Research Site, Haverhill, Massachusetts
  - Research Site, Natick, Massachusetts
  - Research Site, North Dartmouth, Massachusetts
  - Research Site, West Roxbury, Massachusetts
  - Research Site, Whitman, Massachusetts
  - Research Site, Worcester, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Grand Rapids, Michigan
  - Research Site, Lansing, Michigan
  - Research Site, Muskegon, Michigan
  - Research Site, Petoskey, Michigan
  - Research Site, Saginaw, Michigan
  - Research Site, Southfield, Michigan
  - Research Site, Duluth, Minnesota
  - Research Site, Minneapolis, Minnesota
  - Research Site, Saint Louis Park, Minnesota
  - Research Site, Saint Paul, Minnesota
  - Research Site, Columbia, Missouri
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Kalispell, Montana
  - Research Site, Missoula, Montana
  - Research Site, Grand Island, Nebraska
  - Research Site, Lincoln, Nebraska
  - Research Site, Lebanon, New Hampshire
  - Research Site, Hackensack, New Jersey
  - Research Site, Morristown, New Jersey
  - Research Site, Newark, New Jersey
  - Research Site, Summit, New Jersey
  - Research Site, Westwood, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Buffalo, New York
  - Research Site, Cortlandt Manor, New York
  - Research Site, Flushing, New York
  - Research Site, Garden City, New York
  - Research Site, Johnson City, New York
  - Research Site, Kingston, New York
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, Staten Island, New York
  - Research Site, Syracuse, New York
  - Research Site, The Bronx, New York
  - Research Site, Troy, New York
  - Research Site, West Islip, New York
  - Research Site, Williamsville, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Burlington, North Carolina
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Gastonia, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, New Bern, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Akron, Ohio
  - Research Site, Canton, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Garfield Heights, Ohio
  - Research Site, Mayfield Heights, Ohio
  - Research Site, Sandusky, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Tulsa, Oklahoma
  - Research Site, Bend, Oregon
  - Research Site, Hillsboro, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Allentown, Pennsylvania
  - Research Site, Hershey, Pennsylvania
  - Research Site, Lancaster, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Sayre, Pennsylvania
  - Research Site, Wyomissing, Pennsylvania
  - Research Site, Pawtucket, Rhode Island
  - Research Site, Anderson, South Carolina
  - Research Site, Charleston, South Carolina
  - Research Site, Columbia, South Carolina
  - Research Site, Orangeburg, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Chattanooga, Tennessee
  - Research Site, Germantown, Tennessee
  - Research Site, Jackson, Tennessee
  - Research Site, Memphis, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Tullahoma, Tennessee
  - Research Site, Beaumont, Texas
  - Research Site, Dallas, Texas
  - Research Site, Galveston, Texas
  - Research Site, Houston, Texas
  - Research Site, Lubbock, Texas
  - Research Site, Odessa, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Tyler, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Annandale, Virginia
  - Research Site, Midlothian, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Roanoke, Virginia
  - Research Site, Bellingham, Washington
  - Research Site, Kirkland, Washington
  - Research Site, Seattle, Washington
  - Research Site, Tacoma, Washington
  - Research Site, Beloit, Wisconsin
  - Research Site, Madison, Wisconsin
  - Research Site, Milwaukee, Wisconsin
- Argentina (20):
  - Research Site, Adrogué, Buenos Aires
  - Research Site, Bahía Blanca, Buenos Aires
  - Research Site, Capital Federal, Buenos Aires
  - Research Site, Ciudad AutÃ³noma de Buenos Aires, Buenos Aires
  - Research Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Research Site, Coronel Suárez, Buenos Aires
  - Research Site, La Plata, Buenos Aires
  - Research Site, Mar del Plata, Buenos Aires
  - Research Site, Quilmes, Buenos Aires
  - Research Site, San Martín, Buenos Aires
  - Research Site, Córdoba, CÃ³rdoba
  - Research Site, Cipolletti, RÃ-o Negro
  - Research Site, Rosario, Santa Fe Province
  - Research Site, Buenos Aires
  - Research Site, Capital Federal
  - Research Site, Corrientes
  - Research Site, Córdoba
  - Research Site, Mendoza
  - Research Site, Salta
  - Research Site, Santa Fe
- Australia (15):
  - Research Site, Camperdown, New South Wales
  - Research Site, Coffs Harbour, New South Wales
  - Research Site, Concord, New South Wales
  - Research Site, Gosford, New South Wales
  - Research Site, New Lambton Heights, New South Wales
  - Research Site, Randwick, New South Wales
  - Research Site, Chermside, Queensland
  - Research Site, Kippa-Ring, Queensland
  - Research Site, Woolloongabba, Queensland
  - Research Site, Bedford Park, South Australia
  - Research Site, Geelong, Victoria
  - Research Site, Heidelberg, Victoria
  - Research Site, Parkville, Victoria
  - Research Site, Prahran, Victoria
  - Research Site, Nedlands, Western Australia
- Austria (5):
  - Research Site, Innsbruck
  - Research Site, Linz
  - Research Site, Salzburg
  - Research Site, Vienna
  - Research Site, Wels
- Belgium (12):
  - Research Site, Aalst
  - Research Site, Antwerp
  - Research Site, Bonheiden
  - Research Site, Bruges
  - Research Site, Brussels
  - Research Site, Genk
  - Research Site, Ghent
  - Research Site, Hasselt
  - Research Site, Huy
  - Research Site, Leuven
  - Research Site, Roeselare
  - Research Site, Turnhout
- Brazil (13):
  - Research Site, Fortaleza, CearÃ¡
  - Research Site, Salvador, Estado de Bahia
  - Research Site, Goiânia, GoiÃ¡s
  - Research Site, Belo Horizonte, Minas Gerais
  - Research Site, Curitiba, ParanÃ¡
  - Research Site, Recife, Pernambuco
  - Research Site, Porto Alegre, Rio Grande do Sul
  - Research Site, Campinas, SÃ£o Paulo
  - Research Site, RiberÃ£o Preto, SÃ£o Paulo
  - Research Site, São Paulo, SÃ£o Paulo
  - Research Site, SÃ£o JosÃ© Do Rio Preto, SÃ£o Paulo
  - Research Site, SÃ£o Paulo, SÃ£o Paulo
  - Research Site, Rio de Janeiro
- Bulgaria (8):
  - Research Site, Dimitrovgrad
  - Research Site, Haskovo
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Rousse
  - Research Site, Sofia
  - Research Site, Varna
  - Research Site, Veliko Tarnovo
- Canada (22):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Campbell River, British Columbia
  - Research Site, Surrey, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Halifax, Nova Scotia
  - Research Site, Ajax, Ontario
  - Research Site, Cambridge, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Kingston, Ontario
  - Research Site, London, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, North York, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Scarborough Village, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Sherbrooke, Quebec
  - Research Site, St-JÃ©rÃ´me, Quebec
  - Research Site, Regina, Saskatchewan
  - Research Site, Saskatoon, Saskatchewan
- Chile (7):
  - Research Site, Rancagua, Cachapoal
  - Research Site, La Serena, Elqui
  - Research Site, San Miguel, Santiago Metropolitan
  - Research Site, Osorno
  - Research Site, Santiago
  - Research Site, Temuco
  - Research Site, Viña del Mar
- Czechia (10):
  - Research Site, Benešov
  - Research Site, Brno
  - Research Site, České Budějovice
  - Research Site, Jihlava
  - Research Site, Karlovy Vary
  - Research Site, Pardubice
  - Research Site, Prague
  - Research Site, Příbram
  - Research Site, Tábor
  - Research Site, Ústí nad Labem
- Denmark (14):
  - Research Site, Fredericia
  - Research Site, Frederiksberg
  - Research Site, Frederikshavn
  - Research Site, Glostrup Municipality
  - Research Site, Hellerup
  - Research Site, Herlev
  - Research Site, Horsens
  - Research Site, Hvidovre
  - Research Site, KÃ¸benhavn Ã˜
  - Research Site, KÃ¸benhavn S
  - Research Site, KÃ¸ge
  - Research Site, Odense
  - Research Site, Roskilde
  - Research Site, Svendborg
- Estonia (2):
  - Research Site, PÃ¤rnu
  - Research Site, Tallinn
- Finland (4):
  - Research Site, Espoo
  - Research Site, Helsinki
  - Research Site, Lahti
  - Research Site, Seinäjoki
- France (19):
  - Research Site, Bron
  - Research Site, Caen
  - Research Site, Cholet
  - Research Site, CrÃ©teil Cedex
  - Research Site, Douai
  - Research Site, Grenoble
  - Research Site, Lille
  - Research Site, Montfermeil
  - Research Site, Montpellier
  - Research Site, Nice
  - Research Site, Paris
  - Research Site, Pessac
  - Research Site, Poitiers
  - Research Site, Pontoise
  - Research Site, Rouen
  - Research Site, Saint-Herblain
  - Research Site, Strasbourg
  - Research Site, Toulouse
  - Research Site, Vandœuvre-lès-Nancy
- Germany (21):
  - Research Site, Bad TÃ¶lz
  - Research Site, Berlin
  - Research Site, Bochum
  - Research Site, Bremen
  - Research Site, Frankfurt
  - Research Site, GÃ¶ttingen
  - Research Site, GeorgsmarienhÃ¼tte
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Heidelberg
  - Research Site, Homburg
  - Research Site, Ingelheim
  - Research Site, KÃ¶ln
  - Research Site, Lahr
  - Research Site, Leipzig
  - Research Site, Mainz
  - Research Site, Marburg
  - Research Site, NÃ¼rnberg
  - Research Site, Schwedt
  - Research Site, Stuttgart
  - Research Site, Witten
- Hong Kong (2):
  - Research Site, Hong Kong
  - Research Site, New Territories
- Hungary (13):
  - Research Site, Békéscsaba
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Győr
  - Research Site, Kalocsa
  - Research Site, Kecskemét
  - Research Site, Sopron
  - Research Site, Szeged
  - Research Site, Szekszárd
  - Research Site, Székesfehérvár
  - Research Site, Szolnok
  - Research Site, Veszprém
  - Research Site, Zalaegerszeg
- India (16):
  - Research Site, Hyderabad, Andhra Pradesh
  - Research Site, Ahmedabad, Gujarat
  - Research Site, Gurgaon, Haryana
  - Research Site, Bangalore, Karnataka
  - Research Site, Mumbai, Maharashtra
  - Research Site, Nagpur, Maharashtra
  - Research Site, Nashik, Maharashtra
  - Research Site, Pune, Maharashtra
  - Research Site, New Delhi, National Capital Territory of Delhi
  - Research Site, Ludhiana, Punjab
  - Research Site, Bikaner, Rajasthan
  - Research Site, Chennai, Tamil Nadu
  - Research Site, Coimbatore, Tamil Nadu
  - Research Site, Madurai, Tamil Nadu
  - Research Site, Lucknow, Uttar Pradesh
  - Research Site, Mumbai
- Israel (11):
  - Research Site, Askelon
  - Research Site, Beer Yaakov
  - Research Site, Beersheba
  - Research Site, Giv‘atayim
  - Research Site, Hadera
  - Research Site, Haifa
  - Research Site, Holon
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Safed
  - Research Site, Tel Aviv
- Italy (20):
  - Research Site, Arezzo
  - Research Site, Bergamo
  - Research Site, Cesenatico (FC)
  - Research Site, Cetraro CS
  - Research Site, Cortona AR
  - Research Site, Eboli
  - Research Site, Ferrara
  - Research Site, ForlÃ¬
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Oliveto Citra SA
  - Research Site, Palermo
  - Research Site, Palmanova UD
  - Research Site, Pavia
  - Research Site, Roma
  - Research Site, Rozzano MI
  - Research Site, San Bonifacio VR
  - Research Site, Torino
  - Research Site, Trento
  - Research Site, Udine
- Latvia (4):
  - Research Site, Daugavpils
  - Research Site, Ogre
  - Research Site, Rēzekne
  - Research Site, Riga
- Lithuania (5):
  - Research Site, Alytus
  - Research Site, Kaunas
  - Research Site, Klaipėda
  - Research Site, Šiauliai
  - Research Site, Vilnius
- Mexico (9):
  - Research Site, Guadajalara, Jalisco
  - Research Site, Guadalajara, Jalisco
  - Research Site, Mexico City, Mexico City
  - Research Site, Monterrey, Nuevo LeÃ³n
  - Research Site, San Luis Potosí City, San Luis PotosÃ-
  - Research Site, Xalapa, Veracruz
  - Research Site, Mérida, YucatÃ¡n
  - Research Site, Baja California
  - Research Site, Distrito Federal
- Netherlands (25):
  - Research Site, 's-Hertogenbosch
  - Research Site, Alkmaar
  - Research Site, Almelo
  - Research Site, Amsterdam
  - Research Site, Arnhem
  - Research Site, Assen
  - Research Site, Blaricum
  - Research Site, Breda
  - Research Site, Delft
  - Research Site, Deventer
  - Research Site, Eindhoven
  - Research Site, Enschede
  - Research Site, Groningen
  - Research Site, Haarlem
  - Research Site, Harderwijk
  - Research Site, Heerlen
  - Research Site, Hilversum
  - Research Site, Hoorn
  - Research Site, Nijmegen
  - Research Site, Rotterdam
  - Research Site, Sneek
  - Research Site, The Hague
  - Research Site, Tiel
  - Research Site, Tilburg
  - Research Site, Zwijndrecht
- Norway (7):
  - Research Site, Arendal
  - Research Site, Ã…lesund
  - Research Site, Gjettum
  - Research Site, Kristiansand
  - Research Site, Oslo
  - Research Site, Skien
  - Research Site, Stavanger
- Poland (13):
  - Research Site, Bialystok
  - Research Site, Gdansk
  - Research Site, Gdynia
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Lublin
  - Research Site, Stalowa Wola
  - Research Site, Tarnów
  - Research Site, Warsaw
  - Research Site, Wałbrzych
  - Research Site, Wroclaw
  - Research Site, Zabrze
  - Research Site, Zielona Góra
- Portugal (3):
  - Research Site, Coimbra
  - Research Site, Faro
  - Research Site, Lisbon
- Research Site, San Juan, Puerto Rico
- Romania (9):
  - Research Site, Arad
  - Research Site, Bacau
  - Research Site, Brasov
  - Research Site, Bucharest
  - Research Site, Iași
  - Research Site, Oradea
  - Research Site, Sibiu
  - Research Site, Târgu Mureş
  - Research Site, Timișoara
- Russia (3):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, Volgograd
- Slovakia (8):
  - Research Site, Bardejov
  - Research Site, Bratislava
  - Research Site, Košice
  - Research Site, Levice
  - Research Site, Lučenec
  - Research Site, Nitra
  - Research Site, Prešov
  - Research Site, Žilina
- South Africa (9):
  - Research Site, Boksburg, Gauteng
  - Research Site, Johannesburg, Gauteng
  - Research Site, Pretoria, Gauteng
  - Research Site, Soweto, Gauteng
  - Research Site, Durban, KwaZulu-Natal
  - Research Site, Parow, Western Cape
  - Research Site, Somerset West, Western Cape
  - Research Site, Worcester, Western Cape
  - Research Site, Cape Town
- Spain (15):
  - Research Site, CÃ³rdoba, AndalucÃ-a
  - Research Site, Granada, AndalucÃ-a
  - Research Site, MÃ¡laga, AndalucÃ-a
  - Research Site, Santander, Cantabria
  - Research Site, Badalona, CataluÃ±a
  - Research Site, Barcelona, CataluÃ±a
  - Research Site, Sabadell, CataluÃ±a
  - Research Site, Tarragona, CataluÃ±a
  - Research Site, Santiago de Compostela, Galicia
  - Research Site, Majadhonda, Madrid
  - Research Site, El Palmar, Murcia
  - Research Site, Galdakao, PaÃ-s Vasco
  - Research Site, Oviedo, Principality of Asturias
  - Research Site, Valencia, Valencia
  - Research Site, Madrid
- Sweden (10):
  - Research Site, Ã-rebro
  - Research Site, Danderyd
  - Research Site, GÃ¶teborg
  - Research Site, LinkÃ¶ping
  - Research Site, MalmÃ¶
  - Research Site, MÃ¶lndal
  - Research Site, Stockholm
  - Research Site, Sundsvall
  - Research Site, UmeÃ¥
  - Research Site, Uppsala
- Switzerland (2):
  - Research Site, Lugano
  - Research Site, Sankt Gallen
- United Kingdom (20):
  - Research Site, Barnet
  - Research Site, Belfast
  - Research Site, Birmingham
  - Research Site, Bradford
  - Research Site, Bridlington
  - Research Site, Cottingham
  - Research Site, Coventry
  - Research Site, Glasgow
  - Research Site, Harrow
  - Research Site, Kirkcaldy
  - Research Site, Leeds
  - Research Site, Leicester
  - Research Site, Livingston
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Romford
  - Research Site, Stockport
  - Research Site, Worcester
  - Research Site, Worthing
  - Research Site, York

REFERENCES:
- [Background] McMurray JJ, Anand IS, Diaz R, Maggioni AP, O'Connor C, Pfeffer MA, Polu KR, Solomon SD, Sun Y, Swedberg K, Tendera M, van Veldhuisen DJ, Wasserman SM, Young JB; RED-HF Committees and Investigators. Design of the Reduction of Events with Darbepoetin alfa in Heart Failure (RED-HF): a Phase III, anaemia correction, morbidity-mortality trial. Eur J Heart Fail. 2009 Aug;11(8):795-801. doi: 10.1093/eurjhf/hfp098. PMID 19633103
- [Background] Swedberg K, Young JB, Anand IS, Cheng S, Desai AS, Diaz R, Maggioni AP, McMurray JJ, O'Connor C, Pfeffer MA, Solomon SD, Sun Y, Tendera M, van Veldhuisen DJ; RED-HF Committees; RED-HF Investigators. Treatment of anemia with darbepoetin alfa in systolic heart failure. N Engl J Med. 2013 Mar 28;368(13):1210-9. doi: 10.1056/NEJMoa1214865. Epub 2013 Mar 10. PMID 23473338
- [Derived] Chung EY, Palmer SC, Saglimbene VM, Craig JC, Tonelli M, Strippoli GF. Erythropoiesis-stimulating agents for anaemia in adults with chronic kidney disease: a network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 13;2(2):CD010590. doi: 10.1002/14651858.CD010590.pub3. PMID 36791280
- [Derived] Abraityte A, Aukrust P, Kou L, Anand IS, Young J, Mcmurray JJV, van Veldhuisen DJ, Gullestad L, Ueland T. T cell and monocyte/macrophage activation markers associate with adverse outcome, but give limited prognostic value in anemic patients with heart failure: results from RED-HF. Clin Res Cardiol. 2019 Feb;108(2):133-141. doi: 10.1007/s00392-018-1331-2. Epub 2018 Jul 26. PMID 30051179
- [Derived] van der Meer P, Grote Beverborg N, Pfeffer MA, Olson K, Anand IS, Westenbrink BD, McMurray JJV, Swedberg K, Young JB, Solomon SD, van Veldhuisen DJ. Hyporesponsiveness to Darbepoetin Alfa in Patients With Heart Failure and Anemia in the RED-HF Study (Reduction of Events by Darbepoetin Alfa in Heart Failure): Clinical and Prognostic Associations. Circ Heart Fail. 2018 Feb;11(2):e004431. doi: 10.1161/CIRCHEARTFAILURE.117.004431. PMID 29367268
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled 13 June 2006; Last patient enrolled 4 May 2012
Period: Overall Study
Arm/Group | Placebo | Darbepoetin Alfa
Started | 1142 | 1136
Received Investigational Product | 1140 | 1133
Completed | 463 (Participants who completed investigational product) | 484 (Participants who completed investigational product)
Not Completed | 679 | 652
Not completed — Ineligibility determined | 4 | 3
Not completed — Adverse Event | 83 | 65
Not completed — Withdrawal by Subject | 111 | 102
Not completed — Participant request | 65 | 64
Not completed — Physician Decision | 47 | 39
Not completed — Lost to Follow-up | 16 | 22
Not completed — Death | 265 | 281
Not completed — Protocol Violation | 64 | 59
Not completed — Pregnancy | 1 | 0
Not completed — Other | 21 | 14
Not completed — Did not receive investigational product | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Darbepoetin Alfa | Total
Number analyzed (Participants) | 1142 | 1136 | 2278
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.6 (11.3) | 70.0 (11.6) | 69.8 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 486 | 458 | 944
  Male | 656 | 678 | 1334
Race/Ethnicity, Customized [Number; unit: participants]
  White or Caucasian | 768 | 781 | 1549
  Black or African American | 113 | 89 | 202
  Hispanic or Latino | 84 | 98 | 182
  Asian | 162 | 162 | 324
  Japanese | 0 | 1 | 1
  American Indian or Alaska Native | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Other | 12 | 3 | 15
Region [Number; unit: participants]
  North America | 323 | 321 | 644
  Latin America and Asia | 286 | 285 | 571
  Western Europe, Israel, South Africa, Australia | 306 | 303 | 609
  Eastern Europe and Russia | 227 | 227 | 454
Device Usage [Number; unit: participants] — Usage of implantable cardioverter defibrillator / cardiac resynchronization therapy (ICD/CRT)
  participants
    CRT with or without ICD | 143 | 143 | 286
    ICD without CRT | 124 | 122 | 246
    None | 875 | 871 | 1746
Kansas City Cardiomyopathy Questionnaire: Overall Summary Score [Mean (Standard Deviation); unit: units on a scale] — The KCCQ is a patient-reported measure for patients with heart failure. It consists of 23 items, is comprised of 7 clinically relevant scales (Symptom Frequency, Burden and Stability, Physical and Social Limitation, Quality of Life, and Self-Efficacy), and yields 3 summary scores (Clinical Summary, Total Symptom, and Overall Summary Scores). Scores range between 0 and 100, with higher scores indicating better health status (eg, better functioning, quality of life, fewer symptoms). Number of participants with available data = 1106 and 1104 for each treatment group respectively, total = 2210.
  units on a scale | 56.5 (22.5) | 55.8 (22.6) | 56.2 (22.5)
Study Specific Characteristic [Kansas City Cardiomyopathy Questionnaire: Symptom Frequency Scale [Mean (Standard Deviation); unit: units on a scale] — The KCCQ is a patient-reported measure for patients with heart failure. It consists of 23 items, is comprised of 7 clinically relevant scales (Symptom Frequency, Burden and Stability, Physical and Social Limitation, Quality of Life, and Self-Efficacy), and yields 3 summary scores (Clinical Summary, Total Symptom, and Overall Summary Scores). Scores range between 0 and 100, with higher scores indicating better health status (eg, better functioning, quality of life, fewer symptoms). Number of participants with available data = 1106 and 1104 for each treatment group respectively, total = 2210.
  units on a scale | 63.3 (25.2) | 63.1 (25.6) | 63.2 (25.4)

OUTCOME MEASURES:

1. Primary Outcome: Time to All Cause Death or First Hospitalization for Worsening Heart Failure
Description: Time to death from any cause or first hospital admission for worsening heart failure (adjudicated by the Clinical Endpoint Committee), whichever occurred first, estimated by Kaplan-Meier method. Participants not experiencing a qualifying event during the study were censored at their last contact time or the study termination date, whichever occurred first.
Time Frame: From randomization to the end of study; maximum time on study was 73 months
Population: Intent-to-treat (ITT) analysis set, defined as all randomized participants
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo | Darbepoetin Alfa
Number analyzed (Participants) | 1142 | 1136
days | 1260.0 [387.0 to 2176.0] | 1184.0 [445.0 to 2074.0]
Statistical Analysis 1: Comparison: Placebo vs Darbepoetin Alfa; Test type: Superiority or Other; p = 0.871, Stratified Log Rank — Stratification factors are: region and type of device (cardiac resynchronization therapy (CRT) with or without implantable cardioverter defibrillator (ICD), ICD without CRT, or none); Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.90 to 1.13] — The hazard ratio and 95% confidence intervals are from the Cox proportional hazards model adjusted by the stratification factors

2. Secondary Outcome: Time to Death From Any Cause
Description: Time from randomization to death due to any cause, estimated by the Kaplan-Meier method. Participants not experiencing a qualifying event during the study were censored at their last contact time or the study termination date, whichever occurred first.
Time Frame: From randomization to the end of study; maximum time on study was 73 months
Population: Intent-to-treat
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo | Darbepoetin Alfa
Number analyzed (Participants) | 1142 | 1136
days | 1637.0 [766.0 to 2229.0] | 1629.0 [682.0 to 2117.0]
Statistical Analysis 1: Comparison: Placebo vs Darbepoetin Alfa; Test type: Superiority or Other; p = 0.512, Stratified Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.92 to 1.19] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Time to Cardiovascular Death or First Hospital Admission for Worsening Heart Failure
Description: Time to cardiovascular death or first hospital admission for worsening heart failure, whichever occured first, estimated using the Kaplan Meier method. Participants not experiencing a qualifying event during the study were censored at their last contact time or the study termination date, whichever occurred first.
Time Frame: From randomization to the end of study; maximum time on study was 73 months
Population: Intent-to-treat
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo | Darbepoetin Alfa
Number analyzed (Participants) | 1142 | 1136
days | 1414.0 [429.0 to NA] — Could not be calculated due to the low number of events. | 1395.0 [483.0 to NA] — Could not be calculated due to the low number of events.
Statistical Analysis 1: Comparison: Placebo vs Darbepoetin Alfa; Test type: Superiority or Other; p = 0.922, Stratified Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.89 to 1.14] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Change From Baseline to Month 6 in Kansas City Cardiomyopathy Questionnaire (KCCQ) Overall Summary Score
Description: The KCCQ is a disease-specific patient-reported outcomes measure for patients with heart failure. It consists of 23 items, is comprised of 7 clinically relevant scales (Symptom Frequency, Symptom Burden, Symptom Stability, Physical Limitation, Social Limitation, Quality of Life, and Self-Efficacy), and yields 3 summary scores (Clinical Summary, Total Symptom, and Overall Summary Scores). Scale and summary scores range between 0 and 100, with higher scores indicating better health status (eg, better functioning, fewer symptoms, better quality of life). Least squares means were calculated from a mixed effects model estimating treatment effect adjusted for region, type of device, and Baseline KCCQ score.
Time Frame: Baseline and Month 6
Population: Intent-to-treat participants with non-missing change from Baseline to Month 6 in KCCQ score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Darbepoetin Alfa
Number analyzed (Participants) | 929 | 928
units on a scale | 4.48 (0.68) | 6.68 (0.68)
Statistical Analysis 1: Comparison: Placebo vs Darbepoetin Alfa; Test type: Superiority or Other; p = 0.005, Mixed Models Analysis; Mixed effects model estimating treatment effect adjusted for region, type of device, and Baseline KCCQ score; Least Squares Mean Difference = 2.20, 95% CI 2-sided [0.65 to 3.75], Standard Error of Mean 0.79

5. Secondary Outcome: Change From Baseline to Month 6 in KCCQ Symptom Frequency Score
Description: as for outcome 4
Time Frame: Baseline and Month 6
Population: Intent-to-treat participants with non-missing change from Baseline to Month 6 in KCCQ score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Darbepoetin Alfa
Number analyzed (Participants) | 927 | 925
units on a scale | 3.91 (0.76) | 6.20 (0.76)
Statistical Analysis 1: Comparison: Placebo vs Darbepoetin Alfa; Test type: Superiority or Other; p = 0.011, Mixed Models Analysis; Mixed effects model estimating treatment effect adjusted for region, type of device, and Baseline KCCQ score; Least Squares Mean Difference = 2.29, 95% CI 2-sided [0.53 to 4.05], Standard Error of Mean 0.90

ADVERSE EVENTS:
Time Frame: Informed consent to 30 days post treatment. Max time 72 months
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Placebo | Darbepoetin Alfa
Serious Adverse Events (participants affected / at risk) | 741/1140 | 781/1133
Other Adverse Events (participants affected / at risk) | 741/1140 | 710/1133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=1140) | Darbepoetin Alfa (N=1133)
Anaemia (Blood and lymphatic system disorders) | 49 | 23
Anaemia of chronic disease (Blood and lymphatic system disorders) | 0 | 1
Coagulopathy (Blood and lymphatic system disorders) | 1 | 2
Haemolytic anaemia (Blood and lymphatic system disorders) | 2 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 2 | 0
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 2 | 0
Sideroblastic anaemia (Blood and lymphatic system disorders) | 0 | 1
Splenic infarction (Blood and lymphatic system disorders) | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2
Acute coronary syndrome (Cardiac disorders) | 13 | 7
Acute left ventricular failure (Cardiac disorders) | 5 | 5
Acute myocardial infarction (Cardiac disorders) | 21 | 21
Adams-Stokes syndrome (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 27 | 26
Angina unstable (Cardiac disorders) | 26 | 24
Aortic valve incompetence (Cardiac disorders) | 1 | 0
Aortic valve stenosis (Cardiac disorders) | 1 | 1
Arrhythmia (Cardiac disorders) | 10 | 5
Arrhythmia supraventricular (Cardiac disorders) | 2 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 2 | 1
Atrial fibrillation (Cardiac disorders) | 30 | 32
Atrial flutter (Cardiac disorders) | 7 | 3
Atrial tachycardia (Cardiac disorders) | 2 | 2
Atrioventricular block (Cardiac disorders) | 3 | 2
Atrioventricular block complete (Cardiac disorders) | 2 | 2
Bradyarrhythmia (Cardiac disorders) | 1 | 1
Bradycardia (Cardiac disorders) | 4 | 7
Bundle branch block left (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 22 | 31
Cardiac asthma (Cardiac disorders) | 3 | 2
Cardiac discomfort (Cardiac disorders) | 0 | 2
Cardiac disorder (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 273 | 264
Cardiac failure acute (Cardiac disorders) | 16 | 21
Cardiac failure chronic (Cardiac disorders) | 8 | 9
Cardiac failure congestive (Cardiac disorders) | 145 | 126
Cardiac valve disease (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 10 | 14
Cardiogenic shock (Cardiac disorders) | 11 | 17
Cardiomyopathy (Cardiac disorders) | 4 | 2
Cardiopulmonary failure (Cardiac disorders) | 0 | 5
Cardiorenal syndrome (Cardiac disorders) | 1 | 2
Cardiovascular insufficiency (Cardiac disorders) | 0 | 1
Congestive cardiomyopathy (Cardiac disorders) | 2 | 1
Coronary artery disease (Cardiac disorders) | 10 | 4
Coronary artery occlusion (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 4 | 0
Coronary artery thrombosis (Cardiac disorders) | 0 | 2
Hypertensive heart disease (Cardiac disorders) | 1 | 0
Intracardiac thrombus (Cardiac disorders) | 0 | 2
Ischaemic cardiomyopathy (Cardiac disorders) | 5 | 6
Left ventricular dysfunction (Cardiac disorders) | 1 | 3
Left ventricular failure (Cardiac disorders) | 3 | 3
Mitral valve disease (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 4 | 2
Mitral valve stenosis (Cardiac disorders) | 0 | 1
Myocardial fibrosis (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 35 | 36
Myocardial ischaemia (Cardiac disorders) | 5 | 1
Palpitations (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 2
Pericarditis (Cardiac disorders) | 1 | 1
Pulseless electrical activity (Cardiac disorders) | 1 | 2
Right ventricular failure (Cardiac disorders) | 0 | 1
Sick sinus syndrome (Cardiac disorders) | 3 | 1
Sinoatrial block (Cardiac disorders) | 0 | 1
Sinus arrhythmia (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 2
Supraventricular tachycardia (Cardiac disorders) | 2 | 2
Tachyarrhythmia (Cardiac disorders) | 0 | 2
Tachycardia (Cardiac disorders) | 2 | 1
Tachycardia paroxysmal (Cardiac disorders) | 0 | 1
Tricuspid valve incompetence (Cardiac disorders) | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 3 | 6
Ventricular extrasystoles (Cardiac disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 10 | 10
Ventricular tachyarrhythmia (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 24 | 22
Arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 1
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 2 | 1
Ichthyosis (Congenital, familial and genetic disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Hyperparathyroidism (Endocrine disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 3
Cataract diabetic (Eye disorders) | 1 | 0
Diabetic retinopathy (Eye disorders) | 1 | 0
Macular fibrosis (Eye disorders) | 1 | 0
Optic ischaemic neuropathy (Eye disorders) | 0 | 1
Retinal artery occlusion (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 0 | 2
Retinal vein occlusion (Eye disorders) | 1 | 0
Retinopathy (Eye disorders) | 0 | 1
Scleral haemorrhage (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 1
Visual acuity reduced (Eye disorders) | 1 | 0
Vitreous haemorrhage (Eye disorders) | 1 | 0
Abdominal adhesions (Gastrointestinal disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 2 | 2
Abdominal hernia (Gastrointestinal disorders) | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 6 | 13
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 3 | 5
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 1
Abdominal wall haemorrhage (Gastrointestinal disorders) | 0 | 1
Anal polyp (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 3 | 1
Coeliac disease (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 2 | 3
Colitis ischaemic (Gastrointestinal disorders) | 2 | 1
Colonic polyp (Gastrointestinal disorders) | 1 | 0
Colonic stenosis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 8 | 9
Crohn's disease (Gastrointestinal disorders) | 1 | 0
Diabetic gastroparesis (Gastrointestinal disorders) | 1 | 0
Diaphragmatic hernia (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 12 | 12
Diverticular perforation (Gastrointestinal disorders) | 0 | 1
Diverticulum (Gastrointestinal disorders) | 2 | 3
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 2 | 3
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 2
Duodenitis (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 4
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Epigastric discomfort (Gastrointestinal disorders) | 1 | 1
Erosive oesophagitis (Gastrointestinal disorders) | 1 | 0
Faecaloma (Gastrointestinal disorders) | 2 | 1
Functional gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 2 | 3
Gastric ulcer (Gastrointestinal disorders) | 4 | 2
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 2
Gastric ulcer perforation (Gastrointestinal disorders) | 2 | 0
Gastritis (Gastrointestinal disorders) | 4 | 4
Gastritis atrophic (Gastrointestinal disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 0
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 23 | 18
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 2
Gingival bleeding (Gastrointestinal disorders) | 0 | 2
Haematemesis (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 1 | 2
Ileus (Gastrointestinal disorders) | 0 | 3
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1
Inflammatory bowel disease (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 5 | 6
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 2 | 1
Intestinal infarction (Gastrointestinal disorders) | 1 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 1
Intestinal mass (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Intestinal polyp (Gastrointestinal disorders) | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0
Large intestinal ulcer (Gastrointestinal disorders) | 2 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 3
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 5 | 6
Oesophageal achalasia (Gastrointestinal disorders) | 0 | 2
Oesophageal food impaction (Gastrointestinal disorders) | 1 | 0
Oesophageal motility disorder (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 3
Pancreatitis (Gastrointestinal disorders) | 2 | 3
Pancreatitis acute (Gastrointestinal disorders) | 3 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 2
Peptic ulcer (Gastrointestinal disorders) | 0 | 2
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 1 | 1
Poor dental condition (Gastrointestinal disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 4 | 5
Rectal polyp (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 2
Subileus (Gastrointestinal disorders) | 1 | 0
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 0 | 3
Toothache (Gastrointestinal disorders) | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Umbilical hernia, obstructive (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 5
Varices oesophageal (Gastrointestinal disorders) | 0 | 1
Volvulus (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 9 | 9
Adverse drug reaction (General disorders) | 1 | 0
Asthenia (General disorders) | 10 | 8
Cardiac death (General disorders) | 29 | 34
Catheter site haemorrhage (General disorders) | 0 | 1
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 3 | 2
Death (General disorders) | 24 | 18
Device breakage (General disorders) | 0 | 1
Device dislocation (General disorders) | 1 | 1
Device lead damage (General disorders) | 0 | 1
Device malfunction (General disorders) | 8 | 10
Device misuse (General disorders) | 0 | 1
Device stimulation issue (General disorders) | 0 | 1
Drowning (General disorders) | 1 | 0
Fatigue (General disorders) | 2 | 2
General physical health deterioration (General disorders) | 3 | 5
Generalised oedema (General disorders) | 1 | 3
Hernia (General disorders) | 1 | 0
Hyperpyrexia (General disorders) | 0 | 1
Hypothermia (General disorders) | 0 | 1
Impaired healing (General disorders) | 1 | 2
Implant site haematoma (General disorders) | 1 | 2
Implant site pain (General disorders) | 1 | 0
Implant site ulcer (General disorders) | 1 | 0
Inflammation (General disorders) | 0 | 1
Malaise (General disorders) | 2 | 1
Medical device complication (General disorders) | 0 | 4
Medical device pain (General disorders) | 0 | 1
Medical device site reaction (General disorders) | 1 | 0
Multi-organ disorder (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 13 | 5
Necrobiosis (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 27 | 22
Oedema (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 2 | 4
Pain (General disorders) | 1 | 0
Polyp (General disorders) | 0 | 1
Pyrexia (General disorders) | 8 | 8
Sudden cardiac death (General disorders) | 8 | 21
Sudden death (General disorders) | 19 | 11
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Thrombosis in device (General disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Biliary colic (Hepatobiliary disorders) | 0 | 1
Cardiac cirrhosis (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 2 | 0
Cholecystitis (Hepatobiliary disorders) | 3 | 5
Cholecystitis acute (Hepatobiliary disorders) | 3 | 4
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 9
Gallbladder non-functioning (Hepatobiliary disorders) | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1
Hepatic congestion (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hepatic lesion (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 1
Hepatomegaly (Hepatobiliary disorders) | 1 | 0
Hepatorenal failure (Hepatobiliary disorders) | 0 | 1
Liver disorder (Hepatobiliary disorders) | 1 | 0
Heart transplant rejection (Immune system disorders) | 0 | 1
Hypogammaglobulinaemia (Immune system disorders) | 0 | 1
Sarcoidosis (Immune system disorders) | 0 | 1
Abdominal abscess (Infections and infestations) | 0 | 1
Abdominal infection (Infections and infestations) | 1 | 0
Abscess limb (Infections and infestations) | 0 | 3
Abscess neck (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 1
Arthritis bacterial (Infections and infestations) | 2 | 0
Arthritis infective (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 5 | 1
Bacterial infection (Infections and infestations) | 0 | 1
Bacterial sepsis (Infections and infestations) | 0 | 1
Bone tuberculosis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 22 | 12
Bronchitis bacterial (Infections and infestations) | 0 | 1
Bronchopneumonia (Infections and infestations) | 4 | 5
Campylobacter infection (Infections and infestations) | 0 | 2
Catheter site infection (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 16 | 18
Clostridial infection (Infections and infestations) | 1 | 3
Clostridium difficile colitis (Infections and infestations) | 2 | 3
Clostridium difficile sepsis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 0 | 2
Device related infection (Infections and infestations) | 2 | 0
Diabetic foot infection (Infections and infestations) | 1 | 0
Diabetic gangrene (Infections and infestations) | 1 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 4
Endocarditis (Infections and infestations) | 1 | 1
Enterococcal sepsis (Infections and infestations) | 1 | 1
Erysipelas (Infections and infestations) | 3 | 5
Escherichia bacteraemia (Infections and infestations) | 1 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
External ear cellulitis (Infections and infestations) | 1 | 0
Fungaemia (Infections and infestations) | 1 | 0
Gangrene (Infections and infestations) | 4 | 1
Gastroenteritis (Infections and infestations) | 7 | 15
Gastroenteritis clostridial (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 3 | 2
H1N1 influenza (Infections and infestations) | 1 | 0
Helicobacter gastritis (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 2 | 0
Implant site infection (Infections and infestations) | 1 | 1
Incision site infection (Infections and infestations) | 1 | 0
Infected skin ulcer (Infections and infestations) | 0 | 2
Infection (Infections and infestations) | 1 | 3
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 0 | 3
Lobar pneumonia (Infections and infestations) | 8 | 8
Localised infection (Infections and infestations) | 7 | 5
Lower respiratory tract infection (Infections and infestations) | 6 | 7
Lung infection (Infections and infestations) | 1 | 1
Lung infection pseudomonal (Infections and infestations) | 1 | 0
Malaria (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 1
Nosocomial infection (Infections and infestations) | 1 | 0
Oropharyngitis fungal (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 5 | 5
Osteomyelitis chronic (Infections and infestations) | 1 | 0
Otitis externa (Infections and infestations) | 0 | 1
Pelvic abscess (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1
Pneumococcal bacteraemia (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 71 | 86
Pneumonia bacterial (Infections and infestations) | 0 | 1
Pneumonia escherichia (Infections and infestations) | 0 | 1
Pneumonia influenzal (Infections and infestations) | 1 | 0
Pneumonia klebsiella (Infections and infestations) | 1 | 0
Pneumonia staphylococcal (Infections and infestations) | 1 | 0
Post procedural infection (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0
Pseudomonal sepsis (Infections and infestations) | 0 | 1
Pulmonary sepsis (Infections and infestations) | 2 | 0
Pyelonephritis (Infections and infestations) | 1 | 3
Pyelonephritis chronic (Infections and infestations) | 2 | 0
Rectal abscess (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 4 | 10
Respiratory tract infection viral (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 22 | 19
Septic shock (Infections and infestations) | 7 | 21
Sinusitis (Infections and infestations) | 1 | 0
Soft tissue infection (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 1 | 3
Staphylococcal osteomyelitis (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 3 | 0
Streptococcal infection (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0
Superinfection (Infections and infestations) | 0 | 1
Tracheobronchitis (Infections and infestations) | 0 | 1
Tuberculous pleurisy (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 4
Urinary tract infection (Infections and infestations) | 20 | 29
Urosepsis (Infections and infestations) | 9 | 8
Viral infection (Infections and infestations) | 1 | 1
Wound infection (Infections and infestations) | 1 | 0
Wound sepsis (Infections and infestations) | 1 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 2 | 1
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 1
Burns third degree (Injury, poisoning and procedural complications) | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 2
Chest injury (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 1
Confusion postoperative (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1
Cystitis radiation (Injury, poisoning and procedural complications) | 0 | 1
Drug administered at inappropriate site (Injury, poisoning and procedural complications) | 0 | 1
Eschar (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 8 | 16
Femoral neck fracture (Injury, poisoning and procedural complications) | 5 | 7
Femur fracture (Injury, poisoning and procedural complications) | 8 | 8
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 1
Hip fracture (Injury, poisoning and procedural complications) | 18 | 14
Humerus fracture (Injury, poisoning and procedural complications) | 3 | 3
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 4 | 3
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Poisoning (Injury, poisoning and procedural complications) | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 2
Rib fracture (Injury, poisoning and procedural complications) | 1 | 3
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Shunt occlusion (Injury, poisoning and procedural complications) | 0 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 2 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 7 | 2
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 7 | 5
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 3 | 6
Wound (Injury, poisoning and procedural complications) | 1 | 2
Wound necrosis (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 2 | 1
Arteriogram coronary (Investigations) | 1 | 0
Blood glucose decreased (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 0 | 1
Blood potassium increased (Investigations) | 0 | 1
Blood uric acid increased (Investigations) | 1 | 0
C-reactive protein abnormal (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 0 | 2
Cardiac output decreased (Investigations) | 0 | 1
Coagulation time prolonged (Investigations) | 1 | 0
Drug level increased (Investigations) | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 2
Glycosylated haemoglobin increased (Investigations) | 0 | 1
Haemodynamic test abnormal (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 3 | 1
International normalised ratio abnormal (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 4 | 5
Liver function test abnormal (Investigations) | 1 | 0
Occult blood (Investigations) | 1 | 0
Occult blood positive (Investigations) | 1 | 1
Platelet count decreased (Investigations) | 0 | 1
Renal function test abnormal (Investigations) | 0 | 1
Transaminases increased (Investigations) | 1 | 1
Transferrin saturation decreased (Investigations) | 0 | 1
Waist circumference increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 2
Weight increased (Investigations) | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 0 | 1
Calciphylaxis (Metabolism and nutrition disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 5 | 1
Dehydration (Metabolism and nutrition disorders) | 22 | 19
Diabetes mellitus (Metabolism and nutrition disorders) | 9 | 14
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 5 | 6
Diabetic complication (Metabolism and nutrition disorders) | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 2 | 2
Gout (Metabolism and nutrition disorders) | 10 | 5
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 13 | 7
Hyperkalaemia (Metabolism and nutrition disorders) | 15 | 13
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 18 | 16
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 9
Hyponatraemia (Metabolism and nutrition disorders) | 11 | 7
Hypovolaemia (Metabolism and nutrition disorders) | 5 | 6
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 0
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 4
Bone infarction (Musculoskeletal and connective tissue disorders) | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 1
Fracture pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 2 | 0
Lordosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7 | 7
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 3
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Spinal deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 3
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Acute myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bladder transitional cell carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bone cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carcinoid tumour pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 2
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 5
Lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant anorectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 2
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 3
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Tonsillar neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Altered state of consciousness (Nervous system disorders) | 0 | 1
Balance disorder (Nervous system disorders) | 1 | 1
Brain compression (Nervous system disorders) | 0 | 1
Brain oedema (Nervous system disorders) | 0 | 1
Carotid artery occlusion (Nervous system disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 3
Cerebral haematoma (Nervous system disorders) | 2 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 14 | 27
Cerebrovascular insufficiency (Nervous system disorders) | 0 | 1
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 3 | 3
Dementia (Nervous system disorders) | 0 | 2
Dementia Alzheimer's type (Nervous system disorders) | 0 | 1
Diabetic hyperosmolar coma (Nervous system disorders) | 1 | 0
Diabetic neuropathy (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 13 | 10
Dysarthria (Nervous system disorders) | 1 | 1
Encephalopathy (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 1
Extrapyramidal disorder (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 2
Haemorrhagic stroke (Nervous system disorders) | 3 | 2
Headache (Nervous system disorders) | 3 | 2
Hemiparesis (Nervous system disorders) | 2 | 0
Hemiplegia (Nervous system disorders) | 1 | 1
Hepatic encephalopathy (Nervous system disorders) | 1 | 3
Hypoglycaemic coma (Nervous system disorders) | 1 | 1
Hypoglycaemic unconsciousness (Nervous system disorders) | 0 | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 1
Intercostal neuralgia (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 7 | 8
Lethargy (Nervous system disorders) | 0 | 2
Loss of consciousness (Nervous system disorders) | 3 | 6
Lumbar radiculopathy (Nervous system disorders) | 1 | 0
Mental impairment (Nervous system disorders) | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 3 | 1
Nerve compression (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 2 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 9 | 8
Radiculopathy (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 3
Spinal cord compression (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 2 | 2
Syncope (Nervous system disorders) | 29 | 19
Toxic encephalopathy (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 4 | 7
VIIth nerve paralysis (Nervous system disorders) | 2 | 0
Vocal cord paralysis (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 2
Confusional state (Psychiatric disorders) | 5 | 6
Delirium (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 3
Disorientation (Psychiatric disorders) | 1 | 1
Insomnia (Psychiatric disorders) | 2 | 0
Major depression (Psychiatric disorders) | 2 | 0
Mental status changes (Psychiatric disorders) | 3 | 8
Psychiatric symptom (Psychiatric disorders) | 1 | 0
Restlessness (Psychiatric disorders) | 1 | 0
Sopor (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
Acute prerenal failure (Renal and urinary disorders) | 3 | 1
Anuria (Renal and urinary disorders) | 0 | 1
Azotaemia (Renal and urinary disorders) | 5 | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 2
Haematuria (Renal and urinary disorders) | 3 | 4
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Ischaemic nephropathy (Renal and urinary disorders) | 1 | 0
Oliguria (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1
Polyuria (Renal and urinary disorders) | 0 | 1
Renal artery stenosis (Renal and urinary disorders) | 1 | 3
Renal failure (Renal and urinary disorders) | 37 | 41
Renal failure acute (Renal and urinary disorders) | 62 | 58
Renal failure chronic (Renal and urinary disorders) | 20 | 11
Renal impairment (Renal and urinary disorders) | 4 | 9
Renal injury (Renal and urinary disorders) | 1 | 2
Renal mass (Renal and urinary disorders) | 1 | 0
Renal tubular necrosis (Renal and urinary disorders) | 0 | 1
Urethral disorder (Renal and urinary disorders) | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 2 | 0
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 7 | 9
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 2
Breast haematoma (Reproductive system and breast disorders) | 1 | 0
Epididymitis (Reproductive system and breast disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Pelvic floor muscle weakness (Reproductive system and breast disorders) | 1 | 0
Prostatic disorder (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 8 | 5
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8 | 6
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Choking sensation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 42 | 22
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 29 | 27
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 9 | 11
Pleural fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 | 10
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 9 | 11
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 19 | 13
Respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 3
Diabetic foot (Skin and subcutaneous tissue disorders) | 3 | 3
Dry gangrene (Skin and subcutaneous tissue disorders) | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 2
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Skin maceration (Skin and subcutaneous tissue disorders) | 0 | 1
Skin necrosis (Skin and subcutaneous tissue disorders) | 2 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 12 | 5
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Cardiac pacemaker insertion (Surgical and medical procedures) | 2 | 0
Cardiac resynchronisation therapy (Surgical and medical procedures) | 0 | 2
Cardioversion (Surgical and medical procedures) | 3 | 2
Coronary arterial stent insertion (Surgical and medical procedures) | 1 | 0
Gastrostomy (Surgical and medical procedures) | 0 | 1
Haemodialysis (Surgical and medical procedures) | 1 | 1
Implantable defibrillator insertion (Surgical and medical procedures) | 4 | 1
Percutaneous coronary intervention (Surgical and medical procedures) | 0 | 1
Resuscitation (Surgical and medical procedures) | 0 | 2
Therapy regimen changed (Surgical and medical procedures) | 0 | 1
Accelerated hypertension (Vascular disorders) | 2 | 1
Aortic aneurysm rupture (Vascular disorders) | 0 | 1
Aortic arteriosclerosis (Vascular disorders) | 0 | 1
Arterial insufficiency (Vascular disorders) | 0 | 1
Arteriosclerosis (Vascular disorders) | 1 | 1
Artery dissection (Vascular disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 2
Deep vein thrombosis (Vascular disorders) | 5 | 8
Embolism (Vascular disorders) | 1 | 0
Essential hypertension (Vascular disorders) | 1 | 0
Extremity necrosis (Vascular disorders) | 1 | 1
Femoral artery aneurysm (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 6 | 4
Hypertension (Vascular disorders) | 6 | 8
Hypertensive crisis (Vascular disorders) | 4 | 1
Hypertensive emergency (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 24 | 22
Hypovolaemic shock (Vascular disorders) | 0 | 2
Intermittent claudication (Vascular disorders) | 1 | 3
Intra-abdominal haematoma (Vascular disorders) | 0 | 1
Ischaemia (Vascular disorders) | 1 | 1
Lymphoedema (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 4 | 5
Peripheral arterial occlusive disease (Vascular disorders) | 4 | 7
Peripheral artery aneurysm (Vascular disorders) | 1 | 0
Peripheral artery stenosis (Vascular disorders) | 1 | 1
Peripheral artery thrombosis (Vascular disorders) | 1 | 0
Peripheral embolism (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 5 | 5
Peripheral vascular disorder (Vascular disorders) | 4 | 2
Phlebitis (Vascular disorders) | 1 | 0
Phlebitis superficial (Vascular disorders) | 0 | 1
Poor peripheral circulation (Vascular disorders) | 0 | 1
Poor venous access (Vascular disorders) | 0 | 1
Shock (Vascular disorders) | 0 | 1
Shock haemorrhagic (Vascular disorders) | 0 | 1
Steal syndrome (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 2
Varicose vein (Vascular disorders) | 1 | 0
Venous insufficiency (Vascular disorders) | 0 | 2
Venous thrombosis limb (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=1140) | Darbepoetin Alfa (N=1133)
Angina pectoris (Cardiac disorders) | 60 | 52
Cardiac failure (Cardiac disorders) | 92 | 69
Constipation (Gastrointestinal disorders) | 68 | 81
Diarrhoea (Gastrointestinal disorders) | 135 | 148
Nausea (Gastrointestinal disorders) | 75 | 71
Asthenia (General disorders) | 112 | 88
Fatigue (General disorders) | 84 | 86
Oedema peripheral (General disorders) | 118 | 115
Bronchitis (Infections and infestations) | 88 | 99
Influenza (Infections and infestations) | 71 | 61
Nasopharyngitis (Infections and infestations) | 111 | 117
Upper respiratory tract infection (Infections and infestations) | 73 | 95
Urinary tract infection (Infections and infestations) | 71 | 82
Fall (Injury, poisoning and procedural complications) | 68 | 80
Gout (Metabolism and nutrition disorders) | 75 | 71
Arthralgia (Musculoskeletal and connective tissue disorders) | 78 | 101
Back pain (Musculoskeletal and connective tissue disorders) | 87 | 93
Pain in extremity (Musculoskeletal and connective tissue disorders) | 93 | 94
Dizziness (Nervous system disorders) | 143 | 138
Headache (Nervous system disorders) | 69 | 67
Cough (Respiratory, thoracic and mediastinal disorders) | 132 | 126
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 174 | 157
Hypotension (Vascular disorders) | 83 | 73

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results aftercompletion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.